CLINICAL TRIAL: NCT02876263
Title: Noninvasive Neuromonitoring of Surgery of the Thoracic Aorta
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Juhani Akseli Stewart, Doctoral thesis student, University of Helsinki
Other Study IDs: HUS 133/E6/07
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Cardiopulmonary Arrest; Aortic Aneurysm, Thoracic; Aortic Diseases; Coronary Artery Disease
Keywords: aortic diseases; aortic aneurysm; electroencephalography; Near-Infrared spectroscopy; Transcranial Doppler ultrasonography; Cardiopulmonary arrest; Hypothermia, Induced
MeSH Terms: conditions — Heart Arrest; Aortic Aneurysm, Thoracic; Aortic Diseases; Coronary Artery Disease; Aortic Aneurysm; Hypothermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Study group: Elective and emergency surgery for aneurysm or dissections of the ascending aorta, operated under extracorporeal circulation, protective deep therapeutic hypothermia and circulatory arrest.
- On-pump CABG Group: Elective coronary artery bypass grafting (CABG) for coronary heart disease under extracorporeal circulation
- OPCAB Group: Elective coronary artery bypass grafting (CABG) for coronary heart disease with a beating heart

SUMMARY:
The aim of this prospective, explorative study of noninvasive neuromonitoring was to search potential and practical methods associated with neurological outcome in the perioperative and immediate postoperative setting of surgery of the thoracic aorta. These methods include abbreviated EEG monitoring, near-infrared spectroscopy, transcranial Doppler ultrasound and biochemical markers associated with neuronal damage.

DETAILED DESCRIPTION:
For the purpose of this study, 30 patients undergoing aortic surgery via a median sternotomy (n=29; 97%) or left thoracotomy (n=1; 3%) and cardiopulmonary bypass with deep hypothermic cardiac arrest were recruited. All patients were operated under deep hypothermia and circulatory arrest, with optional selective cerebral perfusion during circulatory arrest. Active patient recruitment started from September 2007 and ended in May 2011. All patients were monitored with a bilateral fronto-temporal four channel abbreviated EEG, a bilateral frontal two-channel near-infrared spectroscopy, postoperative transcranial Doppler ultrasound evaluation of median artery circulation and postoperative biochemical neuromarkers. The study montage was set up by a dedicated research nurse, who also performed the transcranial Doppler measurements. The neuromonitoring data were not used at the time to guide therapeutic decisions, with the exception of near-infrared spectroscopy monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective or emergency surgery on the thoracic aorta (study group) or coronary heart disease (control groups)
* Informed consent from patient or next of kin

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years or older) scheduled for elective or emergency surgery on the thoracic aorta (study group) or coronary heart disease (control groups)
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2007-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Neurological outcome | Monitoring period from anesthesia induction to 48 hours after end of surgery
  Permanent neurological damage or death within monitoring period (up to 48 h after surgery)

CONTACTS AND LOCATIONS:
Overall Officials: Ulla-Stina Salminen, MD, PhD, Study Director — Helsinki University Hospital, Department of Cardiac Surgery
Locations (1):
- Helsinki University Central Hospital, Department of Cardiac Surgery, Helsinki, Uudenmaan Lääni, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simmons LE, Riker RR, Prato BS, Fraser GL. Assessing sedation during intensive care unit mechanical ventilation with the Bispectral Index and the Sedation-Agitation Scale. Crit Care Med. 1999 Aug;27(8):1499-504. doi: 10.1097/00003246-199908000-00016. PMID 10470756
- [Background] Frenzel D, Greim CA, Sommer C, Bauerle K, Roewer N. Is the bispectral index appropriate for monitoring the sedation level of mechanically ventilated surgical ICU patients? Intensive Care Med. 2002 Feb;28(2):178-83. doi: 10.1007/s00134-001-1183-4. Epub 2002 Jan 12. PMID 11907661
- [Background] Jobsis FF. Noninvasive, infrared monitoring of cerebral and myocardial oxygen sufficiency and circulatory parameters. Science. 1977 Dec 23;198(4323):1264-7. doi: 10.1126/science.929199.
- [Background] Hongo K, Kobayashi S, Okudera H, Hokama M, Nakagawa F. Noninvasive cerebral optical spectroscopy: depth-resolved measurements of cerebral haemodynamics using indocyanine green. Neurol Res. 1995 Apr;17(2):89-93. doi: 10.1080/01616412.1995.11740293. PMID 7609855
- [Background] Tiainen M, Roine RO, Pettila V, Takkunen O. Serum neuron-specific enolase and S-100B protein in cardiac arrest patients treated with hypothermia. Stroke. 2003 Dec;34(12):2881-6. doi: 10.1161/01.STR.0000103320.90706.35. Epub 2003 Nov 20. PMID 14631087
- [Background] Lewis PM, Smielewski P, Rosenfeld JV, Pickard JD, Czosnyka M. Monitoring of the association between cerebral blood flow velocity and intracranial pressure. Acta Neurochir Suppl. 2012;114:147-51. doi: 10.1007/978-3-7091-0956-4_27. PMID 22327681